CLINICAL TRIAL: NCT03867955
Title: Study of the Link Between the Slope of the Photomotor Reflex and the Depth of Anesthesia. Prospective, Monocentric, Observational Compendium
Brief Title: Study of the Link Between the Slope of the Photomotor Reflex and the Depth of Anesthesia: "ILLUMINANS" Study
Acronym: ILLUMINANS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN372018/CHUSTE
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Neurosurgical Intervention
Keywords: photomotor reflex; depth of anesthesia; AlgiScan™; pupil diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have a neurosurgical intervention: Patients who have a neurosurgical intervention will be included. They will have a collection of datas.
  Interventions: Other: Collection of datas

INTERVENTIONS:
Other: Collection of datas — Collection of datas by videopupillometer results: pupil diameter and variation of the pupillary diameter.

SUMMARY:
Pupillary diameter monitoring is currently used routinely for assessment of the nociception / antinociception balance during surgery.

Pupillary diameter decreases reflexively in response to light flash, called photomotor reflex. The photomotor reflex is described by the latency between the light flash and the beginning of the decay expressed in milliseconds, the slope or decay rate expressed in millimeters per second, and the percentage of variation, corresponding to the ratio between the basal pupil diameter and the minimum diameter reached during the light stimulation.

The AlgiScan™ videopupillometer used includes a device for producing a flash light, designed for this purpose.

It has recently been shown that the slope (or rate) of pupillary diameter decrease during a light flash varies during anesthesia, independently of any nociceptive stimulus.

DETAILED DESCRIPTION:
The hypothesis of this study is the variation of the decay slope of the pupil diameter is proportional to the depth of the anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Majors patients
* Score American Society of Anesthesiologists (ASA) 1 or 2
* Managed in the operating theater of the University Hospital of Saint-Etienne for a neurosurgical intervention.

Exclusion Criteria:

* Single or bilateral eye surgery modifying the possibilities of variation of the pupillary diameter
* Having been asleep under general anesthesia in the 7 days prior to the current surgery
* History of Parkinson's disease, insulin-dependent or non-insulin-dependent diabetes at a dysautonomic stage or chronic alcoholism at a dysautonomous stage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a neurosurgical intervention will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
slope (or rate) of pupil diameter change | Day 0
  To compare the slope (or rate) of pupil diameter change obtained during a standardized 320 Lux light flash and the depth of anesthesia evaluated by the Bispectral Index (BIS™) at different levels of depth of anesthesia.

SECONDARY OUTCOMES:
latency and the amplitude of pupillary diameter reduction | Day 0
  Correlation between the latency and the amplitude of pupillary diameter reduction obtained during a standardized 320 Lux light flash between the basic pupillary diameter, Pupillary Unrest in Ambient Light (PUAL) and between eyeball movements, and depth of anesthesia as assessed by BIS™.

CONTACTS AND LOCATIONS:
Overall Officials: David CHARIER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No